CLINICAL TRIAL: NCT06438224
Title: Clinical Utility of Extracorporeal Shock Wave Therapy in Restoring Hand Function of Patients With Nerve Injury and Hypertrophic Scars Due to Burns
Brief Title: Clinical Utility of ESWT in Restoring Hand Function of Patients With Nerve Injury and Hypertrophic Scars Due to Burns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HangangSHH-18
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hand Injuries; Extracorporeal Shock Wave Therapy; Burns
Keywords: Extracorporeal shock wave therapy; hypertrophic scar; burns; hand function; nerve injury
MeSH Terms: conditions — Hand Injuries; Burns; Cicatrix, Hypertrophic | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: ESWT was conducted using the Duolith SD-1® device (StorzMedical, Tägerwilen, Switzerland), with an electromagnetic cylindrical coil source used to focus the shock wave. ESWT was performed around the primary treatment site, at an intensity of 100 impulses/cm2, an energy flux density (EFD) of 0.05 to 0.30 mJ/mm2, and frequency of 4 Hz. Regarding the volume of treatment, 1000-3000 impulses were administered per session for 12 sessions held at 1-week intervals. As in previous studies, the sham group was treated using an adapter that had the same shape but did not emit any energy
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome measurements and data analyses were performed by a trained and blinded outcome assessor who was not involved in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal shock wave therapy (ESWT) (Experimental): Those in the ESWT group were asked to select the most hypertrophic and retracting scars for treatment. ESWT was conducted using the Duolith SD-1® device (StorzMedical, Tägerwilen, Switzerland), with an electromagnetic cylindrical coil source used to focus the shock wave. ESWT was performed around the primary treatment site, at an intensity of 100 impulses/cm2, an energy flux density (EFD) of 0.05 to 0.30 mJ/mm2, and frequency of 4 Hz. Regarding the volume of treatment, 1000-3000 impulses were administered per session for 12 sessions held at 1-week intervals.
  Interventions: Other: Extracorporeal shock wave therapy (ESWT)
- sham group (Sham Comparator): the sham group was treated using an adapter that had the same shape but did not emit any energy
  Interventions: Other: sham stimulation

INTERVENTIONS:
Other: Extracorporeal shock wave therapy (ESWT) — Those in the ESWT group were asked to select the most hypertrophic and retracting scars for treatment. ESWT was conducted using the Duolith SD-1® device (StorzMedical, Tägerwilen, Switzerland), with an electromagnetic cylindrical coil source used to focus the shock wave. ESWT was performed around the primary treatment site, at an intensity of 100 impulses/cm2, an energy flux density (EFD) of 0.05 to 0.30 mJ/mm2, and frequency of 4 Hz. Regarding the volume of treatment, 1000-3000 impulses were administered per session for 12 sessions held at 1-week intervals.
  Arms: Extracorporeal shock wave therapy (ESWT)
Other: sham stimulation — the sham group was treated using an adapter that had the same shape but did not emit any energy
  Arms: sham group

SUMMARY:
Joint contractures and nerve injuries are common after hand burns. Extracorporeal shock wave therapy (ESWT) is effective not only for the regeneration of various tissues, including scar tissues, but also for reducing pain and pruritus in patients with burns. Researchers have attempted to explore the effects of ESWT on hand dysfunction caused by nerve injury following burns. The investigators planned to evaluate the effects of ESWT (compared to sham stimulation) on hands with nerve injury and hypertrophic scars and thereby on hand function. The ESWT parameters were as follows: energy flux density, 0.05-0.30 mJ/mm2; frequency, 4 Hz; 1000 to 2000 impulses per treatment; and 12 treatments, one/week for 12 weeks. Outcome measures were as follows: 10-point visual analog scale for pain, Jebsen-Taylor hand function test, grip strength, Purdue Pegboard test, ultrasound measurement of scar thickness, and skin characteristics before and immediately after 12 weeks of treatment.

DETAILED DESCRIPTION:
Burns that occur in the hand cause early joint range-of-motion (ROM) limitations and hand muscle weakness that significantly affect quality of life. Hand burns, though restricted to a small total body surface area (TBSA), can have significant functional consequences. Joint contractures and nerve injuries are common after hand burns. Extracorporeal shock wave therapy (ESWT) is effective not only for the regeneration of various tissues, including scar tissues, but also for reducing pain and pruritus in patients with burns.

The investigators have attempted to explore the effects of ESWT on hand dysfunction caused by nerve injury following burns. The investigators planned to evaluate the effects of ESWT (compared to sham stimulation) on hands with nerve injury and hypertrophic scars and thereby on hand function. The ESWT parameters were as follows: energy flux density, 0.05-0.30 mJ/mm2; frequency, 4 Hz; 1000 to 2000 impulses per treatment; and 12 treatments, one/week for 12 weeks. Outcome measures were as follows: 10-point visual analog scale for pain, Jebsen-Taylor hand function test, grip strength, Purdue Pegboard test, ultrasound measurement of scar thickness, and skin characteristics before and immediately after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* had sustained a deep partial-thickness (second-degree) or a full-thickness (third-degree) burn in the right dominant hand, which had been treated with a split-thickness skin graft (STSG) after the thermal injury
* nerve injury to the hand was confirmed by electromyography
* < 6 months prior to the enrollment

Exclusion Criteria:

* musculoskeletal diseases (fracture, amputation, rheumatoid arthritis, and degenerative joint diseases) of the hands
* acute infection
* malignant tumors
* coagulopathy
* pregnancy
* potential for additional skin damage if exposed to ESWT and conventional occupational therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
10-point visual analog scale (VAS) | 12 weeks
  self-reported pain severity, ratings ranging from 0 (no pain) to 10 (unbearable pain

SECONDARY OUTCOMES:
the total active motion (TAM) scoring system | 12 weeks
  range of motion measurement, higher scores indicating better range of motion. For each finger, the maximum angle is 260 degrees and the minimum angle is 260 degrees.
Jebsen-Taylor hand function test (JTT) | 12 weeks
  The JTT consists of seven subtests, each scored on a 0-15-point scale, with higher scores indicating better hand function
Grip and pinch strengths | 12 weeks
  quantified using a hand-held dynamometer (Lafayette Instrument, USA), with higher socres indicating more stronger
Scar thickness | 12 weeks
  quantified using ultrasonography (128 BW1 US system, Medison, Korea)
erythema | 12 weeks
  Mexameter®(MX18, Courage-Khazaka Electronics GmbH, Germany) was used to measure the melanin levels. Higher values indicated darker.
Trans-epidermal water loss (TEWL) | 12 weeks
  measured using a Tewameter® (Courage-Khazaka Electronic GmbH, Germany) to evaluate water evaporation. Higher values indicated skin dryness
pigmentation | 12 weeks
  Mexameter®(MX18, Courage-Khazaka Electronics GmbH, Germany) was used to measure the severity of erythema. Higher values indicated redder skin.

CONTACTS AND LOCATIONS:
Overall Officials: SO YOUNG JOO, Principal Investigator — handgang sacred heart hospital
Locations (1):
- Hangang sacred heart hodpital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thiele S, Thiele R, Gerdesmeyer L. Lateral epicondylitis: This is still a main indication for extracorporeal shockwave therapy. Int J Surg. 2015 Dec;24(Pt B):165-70. doi: 10.1016/j.ijsu.2015.09.034. Epub 2015 Oct 9. PMID 26455532
- [Result] Cui HS, Hong AR, Kim JB, Yu JH, Cho YS, Joo SY, Seo CH. Extracorporeal Shock Wave Therapy Alters the Expression of Fibrosis-Related Molecules in Fibroblast Derived from Human Hypertrophic Scar. Int J Mol Sci. 2018 Jan 2;19(1):124. doi: 10.3390/ijms19010124. PMID 29301325